CLINICAL TRIAL: NCT03431142
Title: Extended Antiplatelet Therapy With Clopidogrel Alone Versus Clopidogrel Plus Aspirin After Completion of 9- to 12-month Dual Antiplatelet Therapy for ACS Patients With Both High Bleeding and Ischemic Risk.
Brief Title: Optimal antiPlatelet Therapy for High Bleeding and Ischemic RISK Patients Trial
Acronym: OPT-BIRISK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Prof., Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOPIL08732
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Prolonged DAPT in ACS Patients With Hisk of Both Ischemic and Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clopidogrel monotherapy (Experimental): On the basis of 9-12 months of DAPT(aspirin+clopidogrel), continue clopidogrel monotherapy in the following 9 months.
  Interventions: Drug: Clopidogrel
- Clopidogrel plus aspirin (Active Comparator): On the basis of 9-12 months of DAPT(aspirin+clopidogrel), continue DAPT (aspirin+clopidogrel) in the following 9 months.
  Interventions: Drug: Clopidogrel+aspirin

INTERVENTIONS:
Drug: Clopidogrel — Additional 9 months of clopidogrel monotherapy after 9-12 months of DAPT (aspirin+clopidogrel)
  Arms: Clopidogrel monotherapy
Drug: Clopidogrel+aspirin — Additional 9 months of clopidogrel plus aspirin after 9-12 months of DAPT (aspirin+clopidogrel)
  Arms: Clopidogrel plus aspirin

SUMMARY:
Current guidelines recommend that patients with ACS undergoing stent implantation might be offered extended DAPT treatment for up to 30 months if necessary.

Therefore, we designed a prospective, multicenter, randomized, placebo-controlled trial among ACS patients with high-risk on ischemic and bleeding who received a new generation of DES and received 9 to 12 months of DAPT, and evaluated whether clopidogrel monotherapy reduce the risk of bleeding compared with clopidogrel plus ASA in the following 9 months and achieved non-inferior outcomes in preventing ischemic risk.

DETAILED DESCRIPTION:
Current guidelines recommend that patients with ACS undergoing stent implantation might be offered extended DAPT treatment for up to 30 months if necessary. For patients with high risk of both ischemic and hemorrhage, despite prolonged use of DAPT may bring antithrombotic benefit, it may also increase the risk of bleeding. There is an urgent need for specific guiding on intensive antiplatelet therapy in this population of patients to reduce the risk of ischemia and to avoid the risk of bleeding.

Previous studies have shown that, after 12 months of DAPT treatment, continuation of clopidogrel monotherapy may further reduce the risk of ischemia and bleeding compared with aspirin. Therefore, we designed a prospective, multicenter, randomized, placebo-controlled trial among ACS patients with high-risk on ischemic and bleeding who received a new generation of DES and received 9 to 12 months of DAPT, and evaluated whether clopidogrel monotherapy reduce the risk of bleeding compared with clopidogrel plus ASA in the following 9 months and achieved non-inferior outcomes in preventing ischemic risk.

ELIGIBILITY:
Inclusion Criteria:

* ACS patients undergoing PCI (New-Generation DES) and finishing 9-12 months of DAPT
* 18 ~ 85 years old adult patients
* Patients under the age of 65 must meet at least one of the following clinical criteria of high bleeding risk and at least one of the following clinical criteria of high ischemic risk; Patients aged 65-75 must meet one of the following clinical criteria of either high bleeding risk or high ischemic risk.

Clinical criteria of high bleeding risk:

* ≥75 years old
* female
* Iron deficiency anemia
* history of stroke (hemorrhagic or ischemic)
* ongoing medical treatment of diabetes (oral hypoglycemic agents or subcutaneous insulin)
* Chronic kidney disease (eGFR <60mL/min or creatinine clearance<60mL/min)

Clinical criteria of high ischemic risk:

* ≥75 years old
* Multiple coronary lesions
* target lesions required for stent of total length> 30mm
* Thrombotic target lesions
* Bifurcation lesions are Medina 0, 1, 1 or 1, 1, and 1, with stents implanted in both main branch and side branch
* Left main coronary artery (≥50%) or proximal LAD (≥70%) lesions
* Calcified plaques requiring endovascular excision
* acute coronary syndrome with troponin positive
* Previous myocardial infarction, ischemic stroke, diagnosed peripheral arterial disease (PAD), or revascularization due to coronary artery disease (CAD) / PAD
* recurrent myocardial infarction, revascularization, stent thrombosis, stroke in the last 9 months
* ongoing medical treatment of diabetes (oral hypoglycemic agents or subcutaneous insulin)
* Chronic kidney disease (eGFR<60 mL/min or creatinine clearance <60 mL/min)

Exclusion Criteria:

* Discontinuation or termination of DAPT treatment during the past 6 months due to adverse events (bleeding or ischemia) or other conditions
* Surgery plan within 90 days
* Coronary Revascularization (Surgical or Intervention) Program within 90 days
* Dialysis-dependent renal failure
* Moderate or severe hepatic insufficiency (2 times the upper limit of normal for ALT or AST)
* Life expectancy <1 year
* Unable or unwilling to provide informed consent
* Women with childbearing potential
* Platelet count <100000/mm3
* Subjects undergoing warfarin or similar anticoagulant therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7758 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical relevant bleeding events | During 9-month follow up
  defined as BARC type 2-5 bleeding events

SECONDARY OUTCOMES:
All bleeding events | During 9-month follow up
  defined all BARC type 1-5 bleeding events
Major adverse cardiovascular and cerebrovascular events(MACCE) | During 9-month follow up
  defined as a composite endpoints of all-cause death, myofarction, stroke and clinically indicated revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — The General Hospital of Northern Theater Command
Locations (103):
- China (103):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Seventh Medical Center of Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital,Capital Medical University, word2, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital,Capital Medical University, word3, Beijing, Beijing Municipality
  - PLA Rocket Force Characteristic Medical Center, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital Army Medical University, Chongqing, Chongqing Municipality
  - Department of Cardiology, Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality
  - University-Town Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Red Cross Hospital, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Fuwai Hospital Chinese Academy Of Medical Sciences, Shenzhen, Shenzhen, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The First Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Bethune International Peace Hospital, Shijiazhuang, Hebei
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Wuhan Union Hospital China, Wuhan, Hubei
  - Tongji Medical College Of Hust, Wuhan, Hubei
  - People's Hospital Of Hunan Province, Changsha, Hunan
  - The Third Xiangya Hospital Of Central South University, Changsha, Hunan
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - HulunBuir People's Hospital, Hulunbuir, Inner Mongolia
  - Inner Mongolia Forestry General Hospital, Hulunbuir, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Nanjing Jinling Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Soochow University, Suzhou, Jiangsu
  - Xuzhou Cancer Hospital, Xuzhou, Jiangsu
  - The Second Affiliated Hospital Of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Bethune Hospital Of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital Of Jilin University, Changchun, Jilin
  - The Second Hospital Of Jilin University, Changchun, Jilin
  - Jilin Central General Hospital, Jilin, Jilin
  - Jilin City Hospital Of Chemical Industry, word1, Jilin, Jilin
  - Jilin City Hospital Of Chemical Industry, word2, Jilin, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Siping First People's Hospital, Siping, Jilin
  - Anshan Center Hospital, Anshan, Liaoning
  - Benxi Central Hospital, Benxi, Liaoning
  - The First Affiliated Hospital Of Dalian Medical University, Dalian, Liaoning
  - The Second Hospital Of Dalian Medical University, Dalian, Liaoning
  - Dalian Friendship Hospital, Dalian, Liaoning
  - Dandong Central Hospital, Dandong, Liaoning
  - The First Affiliated Hospital Of Liaoning University Of Traditional Chinese Medicine, Shenyang, Liaoning
  - The First Hospital Of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The Fourth Affiliated Hospital Of China Medical University, Shenyang, Liaoning
  - The People's Hospital Of Liaoning Province, Shenyang, Liaoning
  - Yingkou Central Hospital, word1, Yingkou, Liaoning
  - Yingkou Central Hospital, word2, Yingkou, Liaoning
  - The First Affiliated Hospital Of Baotou Medical College, Baotou, Neimonggol
  - Baotou City Central Hospital, Baotou, Neimonggol
  - Inner Mongolia People's Hospital, Hohhot, Neimonggol
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Central Hospital Affiliated To Shandong First Medical University, Jinan, Shandong
  - The General Hospital Of Jinan Military Command, Jinan, Shandong
  - Qilu Hospital Of Shandong University, Jinan, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated To Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, word 1, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, word 2, Chengdu, Sichuan
  - The General Hospital Of Western Theater Command PLA, Chengdu, Sichuan
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, word1, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, word2, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - Beijing Chao-Yang Hospital,Capital Medical University, Beijing
  - Beijing Anzhen Hospital,Capital Medical University， word1, Beijing
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University People's Hospital, Beijing
  - The Sixth Medical Center of PLA General Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Tongren Hospital,CMU, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Li J, Wang B, Jing Q, Zeng Y, Hou A, Wang Z, Liu A, Zhang J, Zhang Y, Zhang P, Jiang D, Liu B, Fan J, Zhang J, Li L, Su G, Yang M, Jiang W, Qu P, Zeng H, Li L, Qiu M, Ru L, Chen S, Zhou Y, Qiao S, Stone GW, Angiolillo DJ, Han Y; OPT-BIRISK Investigators. Extended Clopidogrel Monotherapy vs DAPT in Patients With Acute Coronary Syndromes at High Ischemic and Bleeding Risk: The OPT-BIRISK Randomized Clinical Trial. JAMA Cardiol. 2024 Jun 1;9(6):523-531. doi: 10.1001/jamacardio.2024.0534. PMID 38630489
- [Background] Li Y, Jing Q, Wang B, Wang X, Li J, Qiao S, Chen S, Angiolillo DJ, Han Y. Extended antiplatelet therapy with clopidogrel alone versus clopidogrel plus aspirin after completion of 9- to 12-month dual antiplatelet therapy for acute coronary syndrome patients with both high bleeding and ischemic risk. Rationale and design of the OPT-BIRISK double-blinded, placebo-controlled randomized trial. Am Heart J. 2020 Oct;228:1-7. doi: 10.1016/j.ahj.2020.07.005. Epub 2020 Jul 9. PMID 32739652